CLINICAL TRIAL: NCT05676086
Title: Innovative Policies for Improving Citizens' Health and Wellbeing Addressing Indoor and Outdoor Lighting
Brief Title: Population Based Lighting Study on Older Adults
Acronym: ENLIGHTENme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 467-2022-SPER-AUSLBO
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Lightning Strategies on Health; Circadian Rhythms Photoentrainment; Photoentrainment and Sleep; DLMO

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indoor light intervention (Experimental): Persons allocated to the indoor light intervention arm will be given a lamp to be placed at home
  Interventions: Behavioral: indoor light intervention
- control group (Active Comparator): Persons allocated to the control group will receive no indoor light supplementation and will undergo assessment procedures only
  Interventions: Behavioral: no indoor light

INTERVENTIONS:
Behavioral: indoor light intervention — Persons allocated to the indoor light intervention arm will be given a lamp to be placed at home with specific instructions to install it in a room where they spend most of their time, in order to supplement the existing indoor lighting. Thus, all people of the intervention arm will be equipped with the LUMIE Halo lamp. Utilizing both warm-white and cool-white LEDs, Lumie Halo delivers 10,000 lux at 20 cm at maximum brightness in "Day" Mode. The touch slider allows the user to adjust the brightness while mixing the color temperature of the light.
  Arms: indoor light intervention
Behavioral: no indoor light — Persons allocated to the control group will receive no indoor light supplementation and will undergo assessment procedures only. Exposure to the outdoor intervention will be taken into account in the analysis in three ways, (1) by locating the distance between people's home and the modified outdoor light, (2) by a question about the awareness of the change in outdoor light, timing, and duration of exposure and what they think of it, and (3) by recording the amount of light exposure over the 24 hours during two weeks at baseline and after the 1-year light interventions
  Arms: control group

SUMMARY:
The ENLIGHTENme project aims at collecting evidence about the impact of outdoor and indoor lighting on human health and wellbeing through the development and testing of innovative solutions and policies that will also counteract health inequalities in European cities. In particular, through an open-online Urban Lighting and Health Atlas, ENLIGHTENme will collect and systematize existing data and good practices on urban lighting and will perform an accurate analysis on the correlations among health, wellbeing, lighting and socio-economic factors in three pilot cities: Bologna (Italy), Amsterdam (The Netherlands), and Tartu (Estonia).

DETAILED DESCRIPTION:
The ENLIGHTENme project aims at collecting evidence about the impact of outdoor and indoor lighting on human health and wellbeing through the development and testing of innovative solutions and policies that will also counteract health inequalities in European cities. In particular, through an open-online Urban Lighting and Health Atlas, ENLIGHTENme will collect and systematize existing data and good practices on urban lighting and will perform an accurate analysis on the correlations among health, wellbeing, lighting and socio-economic factors in three pilot cities: Bologna (Italy), Amsterdam (The Netherlands), and Tartu (Estonia).

In this context, the ENLIGHTENme project will also include an interventional, multicenter, prospective, randomized, controlled, unblinded trial involving one target district, selected based on its artificial light characteristics, in the urban areas of each of one of the three pilot cities. Within each target district, a random sample of individuals aged 65 years or older (intervention group) will be exposed to modifications in domestic indoor lighting and compared with a control group, living in the same target district, unexposed to domestic electric light modifications. At the same time, in a specific area of the target district, outdoor lighting will be modified by the local municipal authority. The hypothesis to be tested in this study is that light interventions may improve individual physical and mental health by affecting circadian entrainment, sleep pattern, and mood. Thus, the study is aimed at providing evidence whether the planned change in electric light exposure at both urban public outdoor and domestic indoor lighting levels may impact on physical and mental health by improving photo-entrainment of circadian rhythms to the light-dark cycle

ELIGIBILITY:
Inclusion Criteria:

* Living in the three selected cities within the target district chosen for the study
* Women and men
* Age 65 years or older
* Signing informed consent

Exclusion Criteria:

* Lack of or inability to provide informed consent
* Lack of or inability to allow data collection over the course of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
impact of electric light on sleep quality | Basal+14 days
  to evaluate the impact of electric light on sleep quality as measured with the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-reported questionnaire that measures sleep quality over the previous month. A higher score indicates poorer sleep quality, therefore the hypothesis to be tested is that a participant's sleep quality will improve (i.e. PSQI score will decrease) at the end of the light intervention period compared to baseline.

SECONDARY OUTCOMES:
Change in photoentrainment | from baseline and the end of the light intervention period - 52 weeks
  Change in photoentrainment as measured by the phase angle between DLMO and sleep onset between the baseline and the end of the light intervention period
circadian rest-activity measures | from baseline and the end of the light intervention period - 52 weeks
  Change in circadian rest-activity measures (IS, IV and RA) as well as sleep measures (SE and FI) as derived from actigraphic measurements between the baseline and the end of the light intervention period
Change in mental and physical health | from baseline and the end of the light intervention period - 52 weeks
  Change in mental and physical health as measured by validated and self-reported questionnaires between the baseline and the end of the light intervention period
actigraphic and melatonin assays | - 52 weeks
  Correlation between clinical parameters derived from actigraphic and melatonin assays and the polygenic risk score derived from publicly available summary statistics of Genome-Wide Association Studies (GWAS), as well as the mitochondrial DNA (mtDNA) haplotypes

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs - Istituto Delle Scienze Neurologiche, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27386582/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30523327/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29221677/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30674076/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26505992/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28525301/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25780233/
- See also: Related Info — https://ec.europa.eu/eurostat/documents/3217494/10166544/KS-02-19%E2%80%91681-EN-N.pdf/c701972f-6b4e-b432-57d2-91898ca94893
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11701584/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8871772/